CLINICAL TRIAL: NCT02330536
Title: Cardiopulmonary Effects of Intrathoracic Pressure Overshoot During Carbon Dioxide Insufflation in Thoracoscopic Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Daping Hospital and the Research Institute of Surgery of the Third Military Medical University (Other)
Responsible Party: Principal Investigator, Qingxiang Mao, M.D., Daping Hospital and the Research Institute of Surgery of the Third Military Medical University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: QMao
Record Dates: First submitted 2014-12-24; First posted 2015-01-05 (Estimated); Last update posted 2021-02-24 (Actual); Status verified 2021-02

CONDITIONS: Esophageal Neoplasms
Keywords: Circulatory and Respiratory Physiological Phenomena; Thoracoscopy
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Flowrate A (Experimental): insufflation of carbon dioxide at 8L/min, 8mmHg
  Interventions: Device: Insufflation of carbon dioxide (CO2)
- Flowrate B (Experimental): insufflation of carbon dioxide at 20 L/min, 8mmHg
  Interventions: Device: Insufflation of carbon dioxide (CO2)

INTERVENTIONS:
Device: Insufflation of carbon dioxide (CO2) — After patients were positioned, CO2 was insufflated into right pleural cavity at eight or twenty L/min. during video-assisted thoracoscopic surgery, thoracic pressure, hemodynamic and respiratory parameters were recorded.

SUMMARY:
Video-assisted thoracoscopic surgery (VATS) has become a standard technique for addressing all types of thoracic pathology. Insufflation of carbon dioxide (CO2) into the operated chest cavity could increase lung collapse and improve surgical field view. The actual thoracic pressure values may not be identical with the presetting on the insufflator display. This overshoot pressure during VATS may compromise cardiac and pulmonary function. The purpose of this study is to evaluate the effects of intrathoracic pressure overshoot during two-lung ventilation on the hemodynamic and respiratory function and clarify the relative safety of two different techniques of insufflation.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) Physical Status Ⅰ,Ⅱ
* Patients with esophageal carcinoma
* Elective video-assisted thoracic surgery

Exclusion Criteria:

* Allergic to drugs used in the study
* Refusal of VAST
* Arrhythmia or treated with antiarrhythmic drug
* Surgery type were converted to thoracotomy,
* Massive intraoperative blood loss (> 400ml)

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 232 (Actual)
Dates: Start 2014-12; Primary Completion 2020-07 (Actual); Study Completion 2020-07 (Actual)

PRIMARY OUTCOMES:
thoracic pressure overshoot | one hour during CO2 insufflation
  Time and value of thoracic pressure overshoot during CO2 insufflation
Hemodynamic change | one hour during CO2 insufflation
  Hemodynamic changes during each overshoot including Systolic Blood Pressure, Central Venous Pressure and Heart Rate
Respiratory change | one hour during CO2 insufflation
  Respiratory changes during each overshoot including Peak Inspiratory Pressure, Pressure flat, Arterial Oxygen Saturation and End-tidal Carbon dioxide

REFERENCES:
- [Background] Claus CM, Cury Filho AM, Boscardim PC, Andriguetto PC, Loureiro MP, Bonin EA. Thoracoscopic enucleation of esophageal leiomyoma in prone position and single lumen endotracheal intubation. Surg Endosc. 2013 Sep;27(9):3364-9. doi: 10.1007/s00464-013-2918-3. Epub 2013 Apr 3. PMID 23549763
- [Background] El-Dawlatly AA, Al-Dohayan A, Abdel-Meguid ME, Turkistani A, Alotaiby WM, Abdelaziz EM. Variations in dynamic lung compliance during endoscopic thoracic sympathectomy with CO2 insufflation. Clin Auton Res. 2003 Dec;13 Suppl 1:I94-7. doi: 10.1007/s10286-003-1120-4. PMID 14673684
- [Background] Brock H, Rieger R, Gabriel C, Polz W, Moosbauer W, Necek S. Haemodynamic changes during thoracoscopic surgery the effects of one-lung ventilation compared with carbon dioxide insufflation. Anaesthesia. 2000 Jan;55(1):10-6. doi: 10.1046/j.1365-2044.2000.01123.x. PMID 10594427
- [Derived] Ren Y, Zhu X, Yan H, Chen L, Mao Q. Cardiorespiratory impact of intrathoracic pressure overshoot during artificial carbon dioxide pneumothorax: a randomized controlled study. BMC Anesthesiol. 2022 Mar 23;22(1):76. doi: 10.1186/s12871-022-01621-9. PMID 35321653